CLINICAL TRIAL: NCT05153031
Title: Impact of Percutaneous Cholecystostomy in the Management of Acute Cholecystitis: A Retrospective Cohort Study.
Brief Title: Impact of Percutaneous Cholecystostomy in the Management of Acute Cholecystitis.
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Candido Fernando Alcazar-Lopez, Principal Investigator, Hospital General Universitario de Alicante
Other Study IDs: 11/2021
Record Dates: First submitted 2021-11-07; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Acute Cholecystitis; Percutaneous Cholecystostomy
Keywords: Acute Cholecystitis; percutaneous cholecystostomy; laparoscopic cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- lithiasic acute cholecystitis: Acute cholecystitis with the presence of one or more calculi (gallstones) in the gallbladder.
  Interventions: Other: lithiasic
- alithiasic acute cholecystitis: Acute cholecystitis without the presence of one or more calculi (gallstones) in the gallbladder.
- elective cholecystectomy: Elective surgery is surgery that is scheduled in advance because it does not involve a medical emergency.
- emergency cholecystectomy: Emergence surgery
  Interventions: Procedure: Emergency surgery
- management with percutaneous cholecystostomy alone: Patients that didnt recieve cholecystectomy during de whole study
- managemente with surgery: Patients that recieve cholecystectomy during de whole study
  Interventions: Procedure: cholecystectomy

INTERVENTIONS:
Other: lithiasic — Cholelithiasis is the presence of one or more calculi (gallstones) in the gallbladder.
  Groups: lithiasic acute cholecystitis
Procedure: Emergency surgery — Emergency cholecystectomy
  Groups: emergency cholecystectomy
Procedure: cholecystectomy — cholecystectomy
  Groups: managemente with surgery

SUMMARY:
Percutaneous cholecystostomy (PC) is an increasingly performed procedure for acute cholecystitis (AC), safe and less invasive than laparoscopic cholecystectomy, very useful in selected patients (severe comorbidities, not suitable for surgery/general anesthesia,..) The investigators conduct a retrospective observational study. Period: 2016-2021. Inclusion criteria: Patients treated with PC for AC. Tokyo guidelines TG13/18 the investigators algorithm to treat AC.

The characteristics of the sample undergoing Percutaneous Cholecystostomy, main indications, evolution and clinical results were reported in an initial observational study. Subsequently, a retrospective analytical study was designed to compare various cohorts: lithiasic vs alithiasic Acute Cholecystitis, elective vs emergency surgery or management with PC alone.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is the gold standard for the treatment of acute cholecystitis (AC). Percutaneous cholecystostomy (PC) is an increasingly performed procedure for AC, safe and less invasive than LC, very useful in selected patients (severe comorbidities, not suitable for surgery/general anesthesia,..).

The theoretical advantages offered by PC are the rapid resolution of sepsis and the optimal preparation of the patient for elective LC . Its main drawback is the possibility of recurrence of AC or other biliary events while awaiting LC.

Thus, many questions about PC remain unanswered: how should the catheter be handled and removed? When is the best time to perform LC? Should cholecystectomy be offered to all patients after PC? Does PC complicate subsequent cholecystectomy? How good is the adherence to the Tokyo Guidelines in real life? To answer these questions, the investigators devised the present study involving patients undergoing PC at the investigators center.

The inclusion criteria were: patients undergoing PC diagnosed with AC following the TG13 and TG18 diagnostic criteria. The exclusion criteria were: patients undergoing PC for causes other than AC, such as neoplasms, bile duct alterations or non-therapeutic diagnostic purposes; patients who had previously undergone endoscopic drainage.

The characteristics of the sample undergoing PC, main indications, evolution and clinical results were reported in an initial observational study. Subsequently, a retrospective analytical study was designed to compare various cohorts: lithiasic vs alithiasic AC, elective vs emergency surgery or management with PC alone. Patients' main characteristics, associated morbidity (complications according to Clavien-Dindo grade (CD) and 90-day mortality, need for new drain placement, and surgical approach (laparoscopic vs. open) were compared, following the STROCSS 2019 guidelines.

Variables were compiled from a review of the digitized medical histories which included one year of follow-up. The demographic variables studied were age and sex. Functional status was assessed according to the ASA scale and comorbidity using the Charlson Comorbidity Index (CCI). The type of radiological test used in the diagnosis (ultrasound, computed tomography (CT), nuclear magnetic resonance, cholangioresonance or a combination of these) and laboratory tests (C-reactive protein and leukocyte count) were recorded. Marked local inflammation was defined as gangrenous or emphysematous AC, biliary perforation/peritonitis, or perivesical abscess. Each patient was classified according to the TG13/18 severity scale: Grade I (mild), Grade II (moderate) or Grade III (severe). The degree of adherence to the TG13/18 was taken into account in the indication of PC.

The main indications for PC, total length of hospitalization, time from admission to drainage placement, and drainage duration in days were recorded. The procedure was considered successful when the patient did not require a new drain or emergency surgery, did not die due to the infection, and could be discharged from hospital after PC removal. Even though PC is not a surgical intervention, the Clavien-Dindo complication scale was used.

The patients who underwent cholecystectomy and those placed on the surgical waiting list were recorded, as was the type of surgery (emergency vs elective). In the case of emergency surgery the reason for the intervention was also reported. Approach, conversion rate to open surgery, total length of hospitalization, time from PC to cholecystectomy (in days), and finally complications according to the Clavien-Dindo classification were assessed. Ninety-day mortality rates of patients both after PC and after cholecystectomy were recorded, as well as the causes. As regards clinical evolution, readmission rates for biliary causes (AC, biliary colic, choledocholithiasis, cholangitis and/or pancreatitis) and other causes were reported, along with time until readmission and main reason.

After the general assessment (physical examination, complementary tests and clinical status) the surgical team decided whether to proceed with PC or perform emergency surgery. The PC was placed by interventional radiologists. The technique was performed under local anesthesia in aseptic conditions, guided by ultrasound or CT. Ultrasound-guided transhepatic PC using the Seldinger technique was the usual procedure. Prior to removal, a cholangiography was performed through the catheter in order to check its patency and the passage of the contrast into the duodenum. In some cases, the drain was closed for 24-48 hours to assess tolerance before removal.

Emergency cholecystectomy was performed by the oncall surgical team. If a laparoscopic approach was chosen, it was carried out using the French technique, with dissection of Calot's triangle until the Strasberg critical view of safety was achieved. If an open approach was selected or if conversion from laparoscopic surgery proved necessary, it was carried out via right subcostal laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PC diagnosed with AC following the TG13 and TG18 diagnostic criteria

Exclusion Criteria:

* Patients undergoing PC for causes other than AC, such as neoplasms, bile duct alterations or non-therapeutic diagnostic purposes;
* Patients who had previously undergone endoscopic drainage.

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing PC diagnosed with AC following the TG13 and TG18 diagnostic criteria
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
global successful rate | through study completion, an average of 1.5 year
  the patient did not require a new drain or emergency surgery, did not die due to the infection, and could be discharged from hospital after PC removal
90-days mortality | 90 days
complications rate | through study completion, an average of 1.5 year

SECONDARY OUTCOMES:
total length of hospitalization during acute episode | through study completion, an average of 1.5 year
drainage duration | through study completion, an average of 1.5 year
1-year readmission rate due to biliary complications | 1 year
The degree of adherence to treatment algorithm of the Tokyo Guidelines 13/18 in the indication of PC | through study completion, an average of 1.5 year
cholecystectomy rate | through study completion, an average of 1.5 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miura F, Takada T, Strasberg SM, Solomkin JS, Pitt HA, Gouma DJ, Garden OJ, Buchler MW, Yoshida M, Mayumi T, Okamoto K, Gomi H, Kusachi S, Kiriyama S, Yokoe M, Kimura Y, Higuchi R, Yamashita Y, Windsor JA, Tsuyuguchi T, Gabata T, Itoi T, Hata J, Liau KH; Tokyo Guidelines Revision Comittee. TG13 flowchart for the management of acute cholangitis and cholecystitis. J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):47-54. doi: 10.1007/s00534-012-0563-1. PMID 23307003
- [Background] Pisano M, Allievi N, Gurusamy K, Borzellino G, Cimbanassi S, Boerna D, Coccolini F, Tufo A, Di Martino M, Leung J, Sartelli M, Ceresoli M, Maier RV, Poiasina E, De Angelis N, Magnone S, Fugazzola P, Paolillo C, Coimbra R, Di Saverio S, De Simone B, Weber DG, Sakakushev BE, Lucianetti A, Kirkpatrick AW, Fraga GP, Wani I, Biffl WL, Chiara O, Abu-Zidan F, Moore EE, Leppaniemi A, Kluger Y, Catena F, Ansaloni L. 2020 World Society of Emergency Surgery updated guidelines for the diagnosis and treatment of acute calculus cholecystitis. World J Emerg Surg. 2020 Nov 5;15(1):61. doi: 10.1186/s13017-020-00336-x. PMID 33153472
- [Background] Gulaya K, Desai SS, Sato K. Percutaneous Cholecystostomy: Evidence-Based Current Clinical Practice. Semin Intervent Radiol. 2016 Dec;33(4):291-296. doi: 10.1055/s-0036-1592326. PMID 27904248
- [Background] Yokoe M, Takada T, Strasberg SM, Solomkin JS, Mayumi T, Gomi H, Pitt HA, Garden OJ, Kiriyama S, Hata J, Gabata T, Yoshida M, Miura F, Okamoto K, Tsuyuguchi T, Itoi T, Yamashita Y, Dervenis C, Chan AC, Lau WY, Supe AN, Belli G, Hilvano SC, Liau KH, Kim MH, Kim SW, Ker CG; Tokyo Guidelines Revision Committee. TG13 diagnostic criteria and severity grading of acute cholecystitis (with videos). J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):35-46. doi: 10.1007/s00534-012-0568-9. PMID 23340953
- [Background] Yokoe M, Hata J, Takada T, Strasberg SM, Asbun HJ, Wakabayashi G, Kozaka K, Endo I, Deziel DJ, Miura F, Okamoto K, Hwang TL, Huang WS, Ker CG, Chen MF, Han HS, Yoon YS, Choi IS, Yoon DS, Noguchi Y, Shikata S, Ukai T, Higuchi R, Gabata T, Mori Y, Iwashita Y, Hibi T, Jagannath P, Jonas E, Liau KH, Dervenis C, Gouma DJ, Cherqui D, Belli G, Garden OJ, Gimenez ME, de Santibanes E, Suzuki K, Umezawa A, Supe AN, Pitt HA, Singh H, Chan ACW, Lau WY, Teoh AYB, Honda G, Sugioka A, Asai K, Gomi H, Itoi T, Kiriyama S, Yoshida M, Mayumi T, Matsumura N, Tokumura H, Kitano S, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: diagnostic criteria and severity grading of acute cholecystitis (with videos). J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):41-54. doi: 10.1002/jhbp.515. Epub 2018 Jan 9. PMID 29032636
- [Background] Agha R, Abdall-Razak A, Crossley E, Dowlut N, Iosifidis C, Mathew G; STROCSS Group. STROCSS 2019 Guideline: Strengthening the reporting of cohort studies in surgery. Int J Surg. 2019 Dec;72:156-165. doi: 10.1016/j.ijsu.2019.11.002. Epub 2019 Nov 6. PMID 31704426
- [Background] Hendrix JM, Garmon EH. American Society of Anesthesiologists Physical Status Classification System. 2025 Feb 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441940/ PMID 28722969
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Clavien PA, Sanabria JR, Strasberg SM. Proposed classification of complications of surgery with examples of utility in cholecystectomy. Surgery. 1992 May;111(5):518-26. PMID 1598671
- [Derived] Rubio-Garcia JJ, Velilla Vico D, Villodre Tudela C, Irurzun Lopez J, Contreras Padilla D, Alcazar Lopez C, Carbonell Morote S, Ramia-Angel JM. Impact of percutaneous cholecystostomy in the management of acute cholecystitis: a retrospective cohort study at a tertiary center. Updates Surg. 2023 Jun;75(4):905-914. doi: 10.1007/s13304-023-01499-3. Epub 2023 Mar 29. PMID 36991301